CLINICAL TRIAL: NCT06456827
Title: ''Comparative Evaluation of Change in Bite Force and Levels of Bone Turnover Markers CTX and BALP in Hyperdivergent and Hypodivergent Cases During Retention Phases-A Prospective Clinical Trial ''
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Dr Aaliya
Record Dates: First submitted 2024-06-08; First posted 2024-06-13 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-10

CONDITIONS: Relapse; Bite Force; Biomarker
Keywords: CTX and BALP biomarker , Bite force
MeSH Terms: conditions — Recurrence; Xanthomatosis, Cerebrotendinous | interventions — Bite Force

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vertical grower (Other): Patients belonging to group 1 will be patient with vertical growth pattern who have undergone fixed orthodontic cases and are ready for debonding with FMA of 26 0 or more. Begg's Retainer will be formed by conventional method and delivered within 24 hours of debonding. Changes in levels of bone turnover markers CTX-bone resorption and BALP-bone formation using ELISA and compare the bite force
  Interventions: Other: Bite force and Gcf
- Horizontal grower (Other): Patients belonging to group 2 will be patient with horizontal growth pattern who have undergone Fixed orthodontic cases and are ready for debonding with with FMA Of 24 o or less.Changes in levels of bone turnover markers CTX-bone resorption and BALP-bone formation using ELISA and compare the bite force
  Interventions: Other: Bite force and Gcf

INTERVENTIONS:
Other: Bite force and Gcf — change in bite force will be measured by bite force measuring device at, T0(at the time of retainer delivery), T1(1 month of retainer delivery), T2(3 months of retainer delivery) and T3 (6 months of retainer delivery) ,T4 (12 months of retainer delivery) time interval.
  Changes in the following parameters - changes in change in levels of bone turnover markers CTX and BALP using ELISA at T0(at the time of retainer delivery), T1(1 month of retainer delivery), T2(3 months of retainer delivery) and T3 (6 months of retainer delivery) ,T4 (12 months of retainer delivery) time interval

SUMMARY:
Long-term studies have shown that various occlusal changes occur after the active phase of orthodontic treatment. some of these changes are unwanted changes and are considered as relapse The retention appliances are used to maintain the arch dimensions and alignment of the teeth after completion of the orthodontic treatment. One indicator of the functional state and health of the masticatory system is maximum voluntary bite force (MVBF). Its values vary in accordance to the location of measurement (highest at the first molar, lower at the incisors). People with pronounced horizontal craniofacial growth have somewhat higher values of MVBF, and those with vertical growth have lower values than do those with an average growth pattern. Clinical case reports and descriptive histologic data exist suggesting that bone and tooth remodeling persist for extended periods after removal of appliance or deactivation. A reflection of bone remodelling can be found in the gingival crevicular fluid (GCF) of moving teeth, with decrease or increase in the concentration of biomarker. This prompted us to evaluate the expression of variation in bone turnover marker levels (CTX-Bone resorption marker and BALP -Bone formation marker ) during the retention period. The International Osteoporosis Foundation (IOF) and International Federation of Clinical Chemistry (IFCC) have recommended C-terminal telopeptide of type I collagen (CTX) as one of the reference for BTMs. Hence, The present trial will be undertaken to assess the changes and compare if there is any difference in bite force and change in level of bone biomarker biomarker CTX type 1 collagen(C-terminal telopeptide of type I collagen and bone specific alkaline phosphatase(BALP) in post orthodontic treatment hypodivergent and hyperdivergent cases using beggs retainer over 12 months of period of retention.

DETAILED DESCRIPTION:
The proposed study will be a non-pharmacological, two arm parallel, Prospective, single blind clinical trial to evaluate if there is a difference in retentive characteristics of dentition in two group of post orthodontic treatment patients with vertical growth pattern patients in one group and horizontal growth pattern patients in other group of patients. The present study will be conducted in the Department of Orthodontic and Dentofacial Orthopedics, P.G.I.D.S, Pt. B.D Sharma University of health sciences, Rohtak. The study will be carried out after the institutional approval obtained from ethical committee.

Patient will be allocated to two different study group by the investigator. the data analyst will be blinded regarding the intervention group. The sample size for the proposed study was calculated by using the formula. Total sample size = N = 2σ 2 (Zβ + Zα/2) 2 / (difference of mean )2. sample size of 20 patients was calculated by using the above formula at confidence interval 95% with power 99%.

GROUP 1: patient with vertical growth pattern have who had undergone, fixed orthodontic cases having FMA of 26 0 or more for hyperdivergent cases.

GROUP 2 patient with horizontal growth pattern who had undergone , Fixed orthodontic cases having FMA of 24 o or less for hypodivergent cases.

Changes in levels of bone turnover markers CTX-bone resorption and BALP-bone formation using ELISA. These parameters will be charted at T0, T1, T2, T3,T4 for each patient.

T0 - Records will be obtained at the time of retainer delivery T1 - Records will be obtained after 1month of retainer delivery T2 - Records will be obtained after 3 month of retainer delivery T3- Records will be obtained after 6 months of retainer delivery T4- Records will be obtained after 12 months of retainer delivery

Assessment of bite force will be done using bite force measuring device at T0 - Records will be obtained at the time of retainer delivery T1 - Records will be obtained after 1month of retainer delivery T2 - Records will be obtained after3month of retainer delivery T3- Records will be obtained after 6 months of retainer delivery T4- Records will be obtained after 12 months of retainer delivery

ELIGIBILITY:
Inclusion Criteria:

* Non - growing (18-25) patients who had finished Fixed orthodontic cases ( ready for debonding )with FMA of 26 or more for hyperdivergent cases and FMA of 24 or less for hypodivergent cases
* Optimal functional occlusion at end of treatment (PAR score >70%).
* Littles irregularity index (Pre-treatment <6mm in both upper and lower arch).
* Nonsurgical and non-orthopedic patients and non syndromic patients.
* Optimal periodontal condition and Good oral hygiene (probing depth <3mm, gingival index score <1
* Good compliance regarding retainer wear

Exclusion Criteria:

* Subjects with incomplete orthodontic treatment.
* TMJ disorder patients.
* Any systemic disease affecting bone and general growth.
* Patients with incomplete records.
* Patient who fail to follow up or undergo complete treatment.
* Patient with learning difficulties
* Patients having antibiotic therapy within previous 3 months and used anti -inflammatory drugs in the month before the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-25 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
change in bite force will be measured by bite force measuring device | 12 months
  change in bite force will be measured by bite force measuring device at, T0(at the time of retainer delivery), T1(1 month of retainer delivery), T2(3 months of retainer delivery) and T3 (6 months of retainer delivery) ,T4 (12 months of retainer delivery) time interval.

SECONDARY OUTCOMES:
- changes in change in levels of bone turnover markers | 12 months
  Changes in the following parameters - changes in change in levels of bone turnover markers CTX and BALP using ELISA at T0(at the time of retainer delivery), T1(1 month of retainer delivery), T2(3 months of retainer delivery) and T3 (6 months of retainer delivery) ,T4 (12 months of retainer delivery) time interval

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Rekha, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No